CLINICAL TRIAL: NCT01649219
Title: Intensity of Exercise and Glucose Metabolism
Acronym: PreDiabEx
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oulu (Other)
Collaborators: Finnish Diabetes Association (Other); Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 64/2009
Record Dates: First submitted 2012-07-21; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Prediabetes
Keywords: Prediabetes, objectively measured exercise, glucose and lipid metabolism, dose response, muscle metabolism.
MeSH Terms: conditions — Prediabetic State | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention (Experimental): 3-month supervised exercise intervention 3 times per week; 60min per time.
  Interventions: Behavioral: Exercise
- No intervention (No Intervention): Standard couselling at baseline

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise intervention

SUMMARY:
Our aim is to investigate the effects of a 12-week structured aerobic exercise on fasting and 2 h glucose, insulin and lipid concentrations in sedentary overweight subjects in whom impaired fasting glucose and/or impaired glucose tolerance was observed for the first time.

DETAILED DESCRIPTION:
Study type: Interventional

Study design: Randomized

Endpoint classification: Changes in fasting and 2 h glucose, insulin and lipid concentrations

Intervention model: Parallel assignment

Masking: Open label

Primary purpose: Prevention and dose response assessment of exercise on glucose and lipid metabolism

Condition: Prediabetes

Intervention: Supervised exercise - The training sessions of the intervention group are carried out indoors 3 times a week for 3 months and supervised by an exercise instructor and physician. Each session last for 60 min and include a 5-min warm-up and stretching, a 20-min walking at speeds 2-4 km/h depending of the participant's physical condition, a 5-min stretching and balance training, a 20-min walking, and a 10-min stretching and balance training. After 1.5 months the 5-min stretching and balance training between the two 20-min walkings is excluded, and the walking time become 45 min.

No intervention: control group; couseling at baseline. Participants of the control group are advised to continue their usual physical and dietary habits.

Experimental: 1 -supervised exercise intervention. No intervention: 2 - standard counseling at baseline.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes determined by 2 hr oGTT

Exclusion Criteria:

* any functional limitation or chronic disease that might have limited the physical exercise and testing
* vigorous physical activity/exercise as revealed by questionnaire and physician exam

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Glucose and lipid metabolism | 3-month intervention

SECONDARY OUTCOMES:
Changes in muscle metabolism | 3-months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Herzig, MD,PhD, Principal Investigator — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland